CLINICAL TRIAL: NCT06704321
Title: A Parallel, Randomized, Placebo-Controlled, Double-Blinded Clinical Trial of the Effects of TOTUM-448 on Liver Fat Content, Cardiometabolic Risk Factors and Gut Microbiota Among Both Men and Women with MASLD
Brief Title: Effects of TOTUM-448 on Liver Fat Content, Cardiometabolic Risk Factors and Gut Microbiota Among Participants with MASLD
Acronym: CARDIO-LIVER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Valbiotis (Industry)
Collaborators: CHU de Quebec-Universite Laval (Other); Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other); Laval University (Other); Valbiotis Canada inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022-497
Record Dates: First submitted 2024-11-12; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: MASLD; Cardiometabolic risk factors; Dietary supplement; Plant extracts; Polyphenols; Liver fat content; Magnetic Resonance Imaging; Overweight; Obesity; Glucose metabolism; Oral glucose tolerance test; Insulin sensitivity; Insulin secretion; Fibroscan; Health-related quality of Life; Body composition; Liver function
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Overweight; Obesity; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, parallel, placebo-controlled study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TOTUM-448 (Experimental): The experimental active arm will be supplemented with TOTUM-448 twice per day.
  Interventions: Dietary Supplement: TOTUM-448
- Placebo (Placebo Comparator): The placebo comparator arm will be supplemented with a placebo twice per day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: TOTUM-448 — 16 weeks of TOTUM-448 supplementation (4.284g/day corresponding to 8 capsules per day)
  Arms: TOTUM-448
Dietary Supplement: Placebo — 16 weeks of placebo supplementation (8 capsules per day)
  Arms: Placebo

SUMMARY:
This clinical trial aims to investigate the effects of TOTUM-448, a mix of 5 plant extracts and choline, consumed at the daily regimen of two times per day, on liver fat content, cardiometabolic risk factors and gut microbiota among both men and women with MASLD.

ELIGIBILITY:
Main Inclusion Criteria:

* Men and women aged between 18 and 75 years (including ranges);
* CAP Score ≥288dB/m with liver stiffness results <8kPa (corresponding to F0 to F1 fibrosis score) assessed by Fibroscan®;
* BMI ≥25 and <40 kg/m2 and WC thresholds according to the NAFLD Nomenclature consensus group (Rinella. 2023. Hepatology);
* Weight stable within ± 5% in the last three months.

Main Exclusion Criteria:

* Contraindications to MRI, Fibroscan® and DEXA;
* Suffering from a metabolic disorder susceptible to significantly affect glucose metabolism or plasma lipid levels or that might affect the study outcomes according to the investigator;
* Suffering from an uncontrolled arterial hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg);
* With a history of atherosclerotic cardiovascular disease (ASCVD);
* Taking medication which may affect the study outcomes;
* Alcohol consumption over ≥10 drinks/week for women and ≥15 drinks/week for men (women consuming more than 3 drinks/day and men consuming more than 4 drinks/day will also be excluded) or not agreeing to keep their alcohol consumption habits unchanged throughout the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evolution of liver fat content | Baseline (V1) and End of supplementation after 16 weeks of supplementation (V3)
  Liver fat content measured by MRI

SECONDARY OUTCOMES:
Evolution of lipid profile | Baseline (V1), Following 8 weeks of supplementation (V2) and End of supplementation after 16 weeks of supplementation (V3)
  Measurement of standard lipid profile
Evolution of glucose homeostasis | Baseline (V1), Following 8 weeks of supplementation (V2) and End of supplementation after 16 weeks of supplementation (V3)
  Measurement of glucose homeostasis
Evolution of liver health | Screening (V0), Following 8 weeks of supplementation (V2) and End of supplementation after 16 weeks of supplementation (V3)
  Cap score assessed by Fibroscan
Evolution of inflammation | Baseline (V1), Following 8 weeks of supplementation (V2) and End of supplementation after 16 weeks of supplementation (V3)
  Measurement of hs-CRP in mg /L Measurement of IL-6, MCP-1, RANTES in pg/ml
Evolution of anthropometric variables | Baseline (V1), Following 8 weeks of supplementation (V2) and End of supplementation after 16 weeks of supplementation (V3)
  Measurement of BMI in kg/m²
Evolution of body composition | Baseline (V1) and End of supplementation after 16 weeks of supplementation (V3)
  Evolution of body composition (i.e. total and trunk fat mass, total and trunk lean body mass) measured by Dual Energy X-ray Absorptiometry (DEXA)
Evolution of health-related quality of life | Baseline (V1) and End of supplementation after 16 weeks of supplementation (V3)
  Health-related quality of life (HRQoF) assessed by Medical Outcome Study Short Form - 36 (MOS SF-36), a generic tool to measure and compare the HRQoL on study population.
Evolution of hepatic function | Screening (V0), Baseline (V1), Following 8 weeks of supplementation (V2) and End of supplementation after 16 weeks of supplementation (V3)
  Measurement of liver assessment
Evolution of kidney function | Screening (V0), Baseline (V1), Following 8 weeks of supplementation (V2) and End of supplementation after 16 weeks of supplementation (V3)
  Measurement of kidney assessment
Evolution of hemodynamic measurements | Screening (V0), Baseline (V1), Following 8 weeks of supplementation (V2) and End of supplementation after 16 weeks of supplementation (V3)
  Measurement of systolic and diastolic blood pressure in mmHg
Evolution of complete blood count | Screening (V0), Baseline (V1), Following 8 weeks of supplementation (V2) and End of supplementation after 16 weeks of supplementation (V3)
  Measurement of white blood cells, red blood cells, number of platelets, amount of hemoglobin in the blood, hematocrit, mean red blood volume, mean hemoglobin amount per red blood cell, mean amount of hemoglobin relative to the size of the cell per red blood cell
Evolution of thyroid stimulating hormone | Screening (V0), Baseline (V1), Following 8 weeks of supplementation (V2) and End of supplementation after 16 weeks of supplementation (V3)
  Measurement of thyroid stimulating hormone
Evolution of adverse events (TEAE, STEAE, TEAE leading to investigational product discontinuation, TEAR) | Screening (V0), Baseline (V1), Following 8 weeks of supplementation (V2) and End of supplementation after 16 weeks of supplementation (V3)
  Treatment-Emergent Adverse Events (TEAE), Serious-TEAE (STEAE), TEAE leading to investigational product discontinuation, Treatment-Emergent Adverse Reaction (TEAR)

CONTACTS AND LOCATIONS:
Overall Officials: André Marette, PhD, Principal Investigator — Laval University
Locations (1):
- Institut sur la nutrition et les aliments fonctionnels (INAF), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No